CLINICAL TRIAL: NCT02206217
Title: The Clinical Trial of Myopia Control in Schoolchildren Using the Multi-segment (MS) Lens
Brief Title: Myopia Control With the Multi-segment Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hoya Vision Care (Industry)
Responsible Party: Principal Investigator, Carly Lam, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-ZG3B
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single vision spectacle lens (No Intervention): Single vision lens with power for correcting distance refraction.
- Multiple-Segment spectacle lens (Experimental): A multifocal spectacle lens that corrects distance refraction and provides myopic defocus at the same time.
  Interventions: Device: Multiple-Segment spectacle lens

INTERVENTIONS:
Device: Multiple-Segment spectacle lens — A multifocal spectacle lens that corrects distance refraction and provides myopic defocus images simultaneously. The myopic defocus aims at slowing down myopia progression.
  Other Names: MS lens
  Arms: Multiple-Segment spectacle lens

SUMMARY:
The purpose of this study is to determine if the Multiple-Segment (MS) spectacle lens can slow myopia progression in Hong Kong schoolchildren.

MS lens is also called Defocus Incorporated Multiple Segments (DIMS) spectacle lens

DETAILED DESCRIPTION:
MS lens is a novel lens designed in attempt to slow myopia progression. It is a multifocal spectacle lens which corrects distance refractive error and at the same time produces myopic defocus images on the retina for all distances. The myopic defocus aims at slowing down myopia progression. The purpose of this study is to investigate if the MS lens can slow myopia progression in Hong Kong Chinese schoolchildren. The subjects will be randomly assigned to either treatment group (wear MS lenses) or control group (wear ordinary single vision lenses). Their cycloplegic refraction and axial length will be monitored every six months over 2 years. The changes in refractive errors and axial length in two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrolment: 8-13 year
* Spherical equivalent refractions (SER): -1.00 to -5.00 Dioptres (D)
* Astigmatism and anisometropia of 1.50 D or less
* Spectacle corrected monocular logMAR visual acuity: 0 or better
* Parents' understanding and acceptance of random allocation of grouping

Exclusion Criteria:

* any ocular and systemic abnormalities might affect visual functions or refractive development
* prior treatment of myopic control, e.g. drugs, orthokeratology, progressive addition lenses, bifocal lenses, drugs (e.g. atropine), etc.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University; Chi ho To, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Centre for Myopia Research, The Hong Kong Polytechnic University, Hong Kong, China
- Centre for Myopia Research, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lam CSY, Tang WC, Tse DY, Lee RPK, Chun RKM, Hasegawa K, Qi H, Hatanaka T, To CH. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses slow myopia progression: a 2-year randomised clinical trial. Br J Ophthalmol. 2020 Mar;104(3):363-368. doi: 10.1136/bjophthalmol-2018-313739. Epub 2019 May 29. PMID 31142465
- [Derived] Chun RKM, Zhang H, Liu Z, Tse DYY, Zhou Y, Lam CSY, To CH. Defocus incorporated multiple segments (DIMS) spectacle lenses increase the choroidal thickness: a two-year randomized clinical trial. Eye Vis (Lond). 2023 Sep 15;10(1):39. doi: 10.1186/s40662-023-00356-z. PMID 37715201
- [Derived] Lam CSY, Tang WC, Zhang HY, Lee PH, Tse DYY, Qi H, Vlasak N, To CH. Long-term myopia control effect and safety in children wearing DIMS spectacle lenses for 6 years. Sci Rep. 2023 Apr 4;13(1):5475. doi: 10.1038/s41598-023-32700-7. PMID 37015996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Vision Spectacle Lens | Multiple-Segment Spectacle Lens
Started | 90 | 93
Completed | 81 | 79
Not Completed | 9 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vision Spectacle Lens | Multiple-Segment Spectacle Lens | Total
Number analyzed (Participants) | 90 | 93 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.01 (1.44) | 10.19 (1.46) | 10.09 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 50 | 55 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 90 | 93 | 183
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 90 | 93 | 183
cycloplegic spherical equivalent refraction (SER) [Mean (Standard Deviation); unit: Diopters (D)] | -2.69 (0.98) | -2.92 (1.09) | -2.81 (1.01)
Axial length [Mean (Standard Deviation); unit: mm] | 24.62 (0.82) | 24.85 (1.59) | 24.74 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Cycloplegic Refraction Change in SER
Description: Change in cycloplegic SER (in diopter) that was measured using Shin-Nippon NVision-K 5001 autorefractor.
Time Frame: Baseline and 2 years
Population: completed 2-year study
Measure: Mean (Standard Deviation); unit: Diopters (D)
Groups:
- SV Group: single vision spectacle lens
- MS Group: Multi-segment lens (or called DIMS lens)
Arm/Group | SV Group | MS Group
Number analyzed (Participants) | 81 | 79
Diopters (D) | -0.93 (0.58) | -0.38 (0.53)

2. Secondary Outcome: Axial Length
Description: Axial length (mm) was measured after cycloplegia using IOL Master
Time Frame: Baseline and 2 years
Population: completed 2-year study
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SV Group | MS Group
Number analyzed (Participants) | 81 | 79
mm | 0.53 (0.24) | 0.21 (0.22)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Interventions were only spectacles, not drug or surgery. The subjects only wore spectacle lenses and had regular routine eye examination that the particpants rarely had risk of adverse events.
Arm/Group | SV Group | MS Group
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/93
Other Adverse Events (participants affected / at risk) | 0/90 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT02206217/Prot_SAP_000.pdf